CLINICAL TRIAL: NCT05418257
Title: A Study on the Non-face-to-face Care Using the Phone, Such as Counseling and Prescription, Temporarily Permitted During the COVID-19 Pandemic
Brief Title: A Study on Telemedicine Applied to Actual Outpatient Clinic for Epilepsy
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-04-059-001
Record Dates: First submitted 2022-05-17; First posted 2022-06-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-08

CONDITIONS: Epilepsy
Keywords: Telemedicine; Telehealth; Non-face-to-face
MeSH Terms: conditions — Epilepsy | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual-Outpatients with Epilepsy: Patient who received treatment at Samsung Medical Center more than twice for epilepsy
- Tele-Outpatients with Epilepsy: Patient who received telemedicine at the time of recruitment and treatment at Samsung Medical Center more than twice for epilepsy
  Interventions: Other: (exposure) telemedicine

INTERVENTIONS:
Other: (exposure) telemedicine — medical counseling or treatment only using phone
  Groups: Tele-Outpatients with Epilepsy

SUMMARY:
This is an observational study to confirm the non-inferior effectiveness on health outcomes of tele-counseling or tele-prescription, which was the first outpatient system applied to the actual medical sites in Korea during the coronavirus disease 2019 (COVID-19) pandemic. Researchers collect data using electronic medical records and questionnaires to patients and their caregivers who are continuously receiving outpatient treatment for epilepsy at a single center. The results of the study will be presented by comparing the health outcomes between the non-face-to-face care group and the usual care group.

DETAILED DESCRIPTION:
During the COVID-19 pandemic, temporary phone consultations or prescriptions are being conducted at actual medical sites in Korea. Now, interest about non-face-to-face medical care and expectation that this medical service will be available in the post COVID-19 era are increasing.

The aim to study non-inferior effectiveness of health outcomes for epilepsy by comparing non-face-to-face care with usual care. In this observational study, two groups are recruited in a matched pair parallel in 1:2 allocation at single outpatient clinic. And then investigators collect data such as seizure control, adherence to treatment, adverse drugs reactions by using electronic medical records and questionnaires.

Because epilepsy, the target disease of the study, has chronic and recurrent symptoms, it is necessary for patients to visit the hospital regularly to check their condition. However, there are few neurologists in the province who can treat epilepsy. So that Patients and their caregivers spend a lot of time and money traveling long distances to get treatment.

ELIGIBILITY:
Inclusion Criteria:

* Those who have received outpatient treatment for epilepsy at least twice from the Department of Neurology, Department of Pediatrics, Samsung Medical Center as of the date of participation in the study
* Those who have been taking one or more anticonvulsants for 3 months or more as of the date of participation in the study
* Those who have passed more than one month from the date of discharge from the hospital as of the date of participation in the study (However, hospitalization for examination only does not fall under this standard)

Exclusion Criteria:

* Those who have an experience of inpatient treatment within 1 month as of the date of participation in the study (However, hospitalization for examination only is not classified as hospitalization under this standard)
* Those who have a record of visiting the emergency room within 1 month as of the date of participation in the study (However, visits that are not for epilepsy drug control are not classified as emergency room visits according to this standard)
* Those who have been diagnosed with psychogenic non-epileptic seizure (PNES) through electroencephalogram (EEG)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will conduct surveys and observation to evaluate the non-inferior-effectiveness of a telehealth between patients and guardians at the Samsung Medical Center's pediatric hospitalist service.
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Seizure control - 1) Change from baseline seizure frequency at 6 months | both at the beginning of the study (month 0) and at the end of the study (month 6)
  It will be assessed by semi-structured questionnaire and EMR review about categorizing seizure frequency.
  : several times per day, 1~2 times per day, several times per week, 1~2 times per week, several times per month, 1~2 times per month, several times per year
Seizure control - 2) Change from baseline seizure type at 6 months | both at the beginning of the study (month 0) and at the end of the study (month 6)
  It will be collected by participants' free text description and EMR review and then will be categorized to generalized, tonic, atonic, focal, absence and status epilepticus by physicians.
  Successful seizure control is defined as no step up in category of seizure frequency and no manifestation of new-onset generalized, tonic/atonic seizure with fall or status epilepticus during study period.

SECONDARY OUTCOMES:
adherence to treatment - 1) Medication compliance | at the end of the study (month 6)
  Medication compliance will be collected by self-report using Likert scale from 1 (worst) to 5 (best compliance as possible)
adherence to treatment - 2) Outpatient visit compliance | at the end of the study (month 6)
  Outpatient visit compliance will be assessed by counting complete in-person visit or telephone consultation and no-shows.
Change from baseline adverse drugs reactions at 6 months | both at the beginning of the study (month 0) and at the end of the study (month 6)
  comparing change and new development of adverse drugs reactions between telemedicine group and usual care group

OTHER OUTCOMES:
patient reported experience - 1) Reasons for using current care system (in-person versus telemedicine) | both at the beginning of the study (month 0) and at the end of the study (month 6)
  The reasons and obstacles for using current outpatient system will be collected with questionnaire.
patient reported experience - 2) Estimated time for outpatient visit | at the end of the study (month 6)
  The average round-trip time from patient's house to hospital will be collected by questionnaire and then estimated.
patient reported experience - 3) Estimated cost for outpatient visit | at the end of the study (month 6)
  The opportunity cost will be collected by questionnaire and then estimated.
patient reported experience - 4) Participants satisfaction | at the end of the study (month 6)
  The satisfaction and willingness of participant using opposite outpatient system (in-person vs telemedicine) will be assessed by questionnaires.
patient reported experience - 5) Caregiver satisfaction | at the end of the study (month 6)
  The satisfaction and willingness of caregiver using opposite outpatient system (in-person vs telemedicine) will be assessed by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Seuk, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-go, South Korea